CLINICAL TRIAL: NCT02194036
Title: The Effect of Learning Oriented Physiotherapy on Health-Related Functioning and Quality of Life in Patients With Various Anxiety Disorders
Brief Title: Learning Oriented Physiotherapy - a New Approach
Acronym: LOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Health North Trøndelag (Unknown); Health Møre and Romsdal (Unknown); South Coast Hospital Hf Dps Aust-Agder Units Arendal (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/393 (REK)
Record Dates: First submitted 2014-07-14; First posted 2014-07-18 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Agitation; Anxiety; Dizziness; Pain; Numbness; Depression; Fatigue; Sleep Disturbances
Keywords: Ownership of body; Bodily and mental balance; Learning; Body image; Sensations; Expectations
MeSH Terms: conditions — Psychomotor Agitation; Anxiety Disorders; Dizziness; Pain; Hypesthesia; Depression; Fatigue; Parasomnias | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Learning oriented physiotherapy (Experimental): Learning oriented physiotherapy is a treatment approach based on knowledge from neuroscience and particularly aimed to curb physical symptoms and ailments, but also to regain a sense of better physical balance and mental control. Therapy sessions are normally given every 2 weeks with individual homework lessons between. The therapy will last between 6 to 12 months depending on learning process and individual needs.
  Interventions: Behavioral: Learning Oriented Physiotherapy
- Widely Recognized Psychiatric Treatment (Active Comparator): Standard Outpatient Treatment within the Psychiatric clinic
  Interventions: Behavioral: Widely Recognized Psychiatric Treatment

INTERVENTIONS:
Behavioral: Learning Oriented Physiotherapy — Clinical practice based on a new understanding of the neurobiological basis for the interaction between body and mind, the foundation of learning and what is needed to bring about change of behavior.
  Other Names: LOF
  Arms: Learning oriented physiotherapy
Behavioral: Widely Recognized Psychiatric Treatment — Standard recognized psychiatric treatment tailored to individual needs.
  Other Names: CBT; Speech Therapy
  Arms: Widely Recognized Psychiatric Treatment

SUMMARY:
Outpatients that suffer from different anxiety disorders may have physical ailments that negatively affect daily life functioning and quality of life. LOF is a physical therapy approach focusing on the link between bodily and mental balance and through defined, but simple movements, patients are expected to learn how to cope and reduce health complaints.

This study aims to investigate the short- and longterm effect of LOF compared to other standardized psychiatric treatments given in the clinic on levels of anxiety and depression, health related function and quality of life.

ELIGIBILITY:
The study population will be recruited among patients referred to three Norwegian psychiatric outpatient clinics for anxiety-like conditions. The same criteria for inclusion and exclusion will be applied for the experimental and active comparator group.

Inclusion Criteria:

Participants should be

* 18 years or older
* able to read, write and speak Norwegian
* understand the project information and consent

Exclusion Criteria:

Participants should not

* have ongoing substance abuse or addiction.
* be psychotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in Health Related Quality of Life (HRoQL) | From baseline to 6, 12 and 18 months of follow-up
  In this study HRoQL will be measured by the validated EQ5D questionnaire

SECONDARY OUTCOMES:
Changes in Levels of Anxiety and Depression | From baseline to 6, 12 and 18 months of follow-up
  Hospital Anxiety and Depression Scale (HAD) will be used as instrument to assess levels and changes in anxiety and depression over time
  .

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Petter Granan, phD, Study Director — Oslo University Hospital, Department of Pain Medicine
Locations (3):
- Norway (3):
  - Regional Psychiatric Centre Aust-Agder, Arendal, Aust-Agder
  - Psychiatric Clinic, Molde, Møre and Romsdal
  - Psychiatric Clinic, Levanger, North Trøndelag

REFERENCES:
- [Background] Britt Fadnes, Kirsti Leira and Per Brodal. Learning-oriented physiotherapy. Theory and practice. University Press, 2013.
- See also: A website with information about the learning-oriented therapy as a new approach, based on new knowledge in neuroscience — http://www.balansekoden.no